CLINICAL TRIAL: NCT06325501
Title: The Efficacy Of Misoprostol Versus Oxytocin Infusion On Reducing Blood Loss During Abdominal Myomectomy
Brief Title: Misoprostol Versus Oxytocin Infusion On Reducing Blood Loss During Abdominal Myomectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AA-2024-1
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Myoma;Uterus
Keywords: misoprostol; oxytocin; myomectomy; blood loss
MeSH Terms: conditions — Myofibroma; Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- misoprostol (Active Comparator): receiving a preoperative rectal dose of 800 ug of misoprostol half an hour before surgery
  Interventions: Drug: Misoprostol 200mcg Tab
- oxytocin (Active Comparator): After the induction of general anaesthesia (GA), an infusion of 40 IU oxytocin in 500 ml normal saline was started at the rate of 250 ml/hour
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab — receiving a preoperative rectal dose of 800 ug of misoprostol half an hour before surgery
  Other Names: Misotac
  Arms: misoprostol
Drug: Oxytocin — after the induction of general anaesthesia (GA), an infusion of 40 IU oxytocin in 500 ml normal saline was started at the rate of 250 ml/hour
  Other Names: syntocinone
  Arms: oxytocin

SUMMARY:
Uterine leiomyomas, or fibroids, are common benign tumors among women, especially those over 35 years old. They can cause various issues, including heavy menstrual bleeding, anemia, pelvic pain, and pressure symptoms. Surgery is often necessary for symptomatic fibroids, with hysterectomy recommended for women over 40 and myomectomy for those wishing to preserve their uterus. Myomectomy can be performed using different surgical approaches but can be associated with significant morbidity, particularly major blood loss, especially in abdominal myomectomy, where up to 20% of women may require blood transfusion.

Various interventions have been introduced to reduce bleeding during myomectomy, such as tourniquets, bupivacaine plus epinephrine infiltration, vasopressin injection, preoperative GnRH agonist administration, and preoperative ascorbic acid injection. However, these strategies may have complications, be ineffective, expensive, or require extra steps.

Oxytocin, primarily secreted from the pituitary gland, is crucial for uterine contraction during labor and delivery, and is used to prevent postpartum uterine atony and bleeding. However, caution is needed in its use, especially in women with heart disease or hypovolemia.

Misoprostol, a prostaglandin E1 analogue, can reduce bleeding during myomectomy by promoting myometrial contractions and reducing uterine artery blood flow. It can be administered via multiple routes, with rectal administration showing advantages in maintaining high plasma concentrations during surgery. Studies have investigated the effectiveness of single preoperative rectal doses of misoprostol versus preoperative oxytocin in reducing bleeding during abdominal myomectomy.

ELIGIBILITY:
Inclusión Criteria:

patients aged between 20 to 48 years old. BMI less than 35 kg/m2 symptomatic uterine myomas. Intramyometrial myoma staging from (3 to 6) according to FIGO staging through trans vaginal ultrasonography (TVUSG) or magnetic resonance imaging (MRI) according to FIGO classification.

maximum diameter of the largest myoma is 15 cm. Uterine size between 14 to 28 weeks of pregnancy.

Exclusion Criteria:

1. History of previous myomectomy
2. Allergy to Misoprostol, carbetocin, TXA, ethamsylate, Oxytocin, vasopressin, bupivacaine and epinephrine.
3. Hypertension.
4. Cardiac and Pulmonary diseases.
5. Patients who have bleeding disorders.
6. Patients on antiplatelets or anticoagulant before surgery.
7. Anemia (Hb < 10g %).
8. Chronic endocrine or metabolic diseases such as Diabetes.
9. Renal and hepatic impairment.
10. Moderate and morbid Obesity (body mass index > 35 kg/m2).
11. Cases that will require intraoperative conversion of myomectomy to hysterectomy.
12. Intracavitary, submucosal, pedunculated Subserosal and adnexal Myoma FIGO staging 0,1,2,7,8.
13. history of Gynecological infections (PID), history of abdominal infections e.g.: peritonitis, history of any abdominal or pelvic operation for non-obstetric cause.

    -

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 20-48 years old with symptomatic uterine myoma indicating operative management, abnormal uterine bleeding or bulk-related symptoms, females with infertility or recurrent pregnancy loss, pressure symptoms, and large myoma(s).
Enrollment: 56 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
intra-operative blood loss | time of surgery
  which was measured at the end of surgery by calculating the sum of blood in the suction bottle and the blood absorbed in the sponges. Dry sponges were weighed before the surgery and the blood-soaked sponges were weighed at the end of the surgery

SECONDARY OUTCOMES:
blood transfusion | 24 hours
post-operative Hb | 24 hours
total surgery time | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tarek N Anees, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine, Kasr el ainy hospital, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No